CLINICAL TRIAL: NCT06993025
Title: A Phase II, Open-Label, Single-Arm, Single-Center Study of Ivonescimab in Combination With Liposomal Irinotecan and 5-Fluorouracil/Leucovorin in Patients With Potentially Resectable Biliary Tract Malignancies
Brief Title: Ivonescimab in Combination With Liposomal Irinotecan and 5-FU/LV in Potentially Resectable Biliary Tract Malignancies
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EC-2025-004
Record Dates: First submitted 2025-04-16; First posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-04

CONDITIONS: Biliary Tract Cancer
MeSH Terms: conditions — Biliary Tract Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ivonescimab+chemotherpy (Experimental): After signing informed consent, subjects who meet the inclusion criteria following screening will receive Ivonescimab in combination with irinotecan liposome injection and 5-FU/LV, administered every 3 weeks for 3 cycles, followed by scheduled radical surgery.
  Subjects who achieve successful conversion will resume treatment within 8 weeks after surgery and continue with Ivonescimab in combination with irinotecan liposome injection and 5-FU/LV, administered every 3 weeks for 3 cycles. Subsequently, they will receive Ivonescimab monotherapy until 1 year of treatment is completed.
  Dosing Schedule:
  1. Ivonescimab: 20 mg/kg, Day 1, intravenous infusion (ivgtt), every 3 weeks (Q3W).
  2. Irinotecan Liposome: 70 mg/m², Day 1, intravenous infusion (ivgtt), every 3 weeks (Q3W).
  3. Calcium Folinate (LV): 400 mg/m², Day 1, intravenous infusion (ivgtt), every 3 weeks (Q3W).
  4. 5-FU: 2400 mg/m², Day 1, intravenous infusion (ivgtt), every 3 weeks (Q3W).
  Interventions: Drug: Ivonescimab+chemotherapy

INTERVENTIONS:
Drug: Ivonescimab+chemotherapy — Dosing Schedule:
  1. Ivonescimab: 20 mg/kg, Day 1, intravenous infusion (ivgtt), every 3 weeks (Q3W).
  2. Irinotecan Liposome: 70 mg/m², Day 1, intravenous infusion (ivgtt), every 3 weeks (Q3W).
  3. Calcium Folinate (LV): 400 mg/m², Day 1, intravenous infusion (ivgtt), every 3 weeks (Q3W).
  4. 5-FU: 2400 mg/m², Day 1, intravenous infusion (ivgtt), every 3 weeks (Q3W).
  Other Names: Ivonescimab+Liposomal Irinotecan + 5-FU/LV

SUMMARY:
This Phase II, single-arm, single-center study evaluates the conversion to resectability and safety of Ivonescimab combined with liposomal irinotecan and 5-FU/LV in patients with potentially resectable biliary tract malignancies. Eligible patients receive three cycles of the combination therapy every 3 weeks, followed by surgery. Post-surgery, patients resume treatment for three more cycles and then continue with evoracizumab alone for up to 1 year. Safety is monitored through AE and SAE assessments for at least 30 and 90 days post-last dose, respectively. Biomarker exploration is also conducted in consenting patients.

DETAILED DESCRIPTION:
This trial is a prospective, single-arm, single-center Phase II study to evaluate the success, safety, and tolerability of surgical conversion of Ivonescimab in combination with irinotecan liposome injection and 5-FU/LV in patients with potentially resectable biliary malignancies.

The study included a screening period (no more than 28 days after subjects signed informed consent to the first treatment), a treatment period (including in-treatment visits and end-of-treatment visits), and a follow-up period (including safety visits, disease progression visits, and survival visits). After signing the informed consent, the subjects underwent a screening period within 28 days prior to the initial treatment to determine their eligibility for the study.

After the subjects signed the informed consent, the subjects who met the screening criteria were selected to receive Ivonescimab combined with irinotican liposome injection and 5-FU/LV, administered once every 3 weeks, and then given radical surgical treatment at an elective time after 3 cycles.

Successful conversion subjects resumed treatment within 8 weeks after surgery and received Ivonescimab combined with irinotecan liposome injection and 5-FU/LV every 3 weeks, and continued to receive Ivonescimab treatment for 1 year after 3 cycles.

The safety of the medication is evaluated, and depending on the severity of adverse events (AE) that occur and are associated with the drug, the investigator will take measures to ensure the safety of the subject. After the final dosing, each subject will receive at least 30 days of follow-up AE monitoring and at least 90 days of follow-up SAE monitoring to evaluate subsequent safety.

Biomarkers for predictive efficacy will also be explored, biomarker blood and tumor samples will be collected at baseline and during the trial for subjects who have signed up for biomarker sample collection/collection.

Administration regimen:

1. Ivonescimab: 20mg/kg, d1, ivgtt, Q3W
2. Irinotecan liposomes: 70mg/m2, d1, ivgtt, Q3W
3. Calcium folinate 400mg/m2, d1, ivgtt, Q3W 4.5-FU 2400mg/m2, d1, ivgtt, Q3W

ELIGIBILITY:
Inclusion Criteria:

* Patients eligible for inclusion in this study must meet all of the following criteria:

  1. Informed Consent: Able to provide written informed consent and understand and agree to comply with study requirements and the assessment schedule.
  2. Age and Gender: Age ≥18 years and ≤75 years on the day of signing the Informed Consent Form (ICF), male or female.
  3. Disease Status: Potentially resectable, previously untreated biliary tract malignancy confirmed by histological or cytological evidence.
  4. Tumor Assessment: Tumor evaluated by a hepatobiliary surgeon with sufficient objective evidence to determine irresectability.
  5. Performance Status: Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
  6. Life Expectancy: Estimated survival of more than 12 weeks.
  7. Body Weight: Weight >30 kg.
  8. Prior Therapy: No prior anti-tumor therapy, including but not limited to anti-CTLA-4, anti-VEGF, anti-PD-1, anti-PD-L1, or anti-PD-L2 antibodies.
  9. EnEnough Organ Function
  10. Coagulation: Prothrombin time (PT) ≤1.5×ULN, international normalized ratio (INR) ≤1.5×ULN, and activated partial thromboplastin time (aPTT) ≤1.5×ULN.
  11. Blood Pressure: Systolic blood pressure ≤150 mmHg and diastolic blood pressure ≤90 mmHg during the screening period, with or without antihypertensive medication. No changes to antihypertensive therapy within 1 week prior to the first administration of the study drug.
  12. Contraception: Sexually active males and females of childbearing potential (not surgically sterilized) must agree to use a medically accepted method of contraception (e.g., intrauterine device, contraceptive pill, or condom) during the study treatment period and for 6 months after the last dose of study treatment.

      • Females of childbearing potential must have a negative serum β-human chorionic gonadotropin (β-HCG) test within 7 days prior to study enrollment and must not be breastfeeding.
  13. HBV Management: Patients with detectable HBV DNA levels (≥10 IU/mL or above the limit of detection) and HBV infection (defined as positive hepatitis B surface antigen [HBsAg] and/or hepatitis B core antibody [anti-HBc]) must receive antiviral therapy according to clinical practice prior to study treatment to ensure adequate viral suppression. Antiviral therapy must be continued during the study period and for 6 months after the last dose of study treatment. Patients with positive anti-HBc but undetectable HBV DNA (<10 IU/mL or below the limit of detection) do not require antiviral therapy unless HBV DNA exceeds 10 IU/mL or the limit of detection during the study. Patients with active HBV and HCV co-infection (defined by positive anti-HCV antibody) or active HBV and hepatitis D virus co-infection are excluded.
  14. Voluntary Participation: Willing to voluntarily participate in the clinical trial, comply with study visits and procedures, understand the study requirements, and have signed the informed consent form.

Exclusion Criteria:

* Exclusion Criteria for Study Enrollment

Participants with any of the following conditions are not eligible for this study:

1. Presence of unresectable extrahepatic metastases.
2. Prior treatment for cholangiocarcinoma, including chemotherapy, molecularly targeted agents, traditional Chinese medicine with antitumor properties, radiotherapy, or interventional therapy (excluding percutaneous transhepatic cholangial drainage [PTCD] or common bile duct stenting). This also includes prior immunotherapy for cholangiocarcinoma.
3. History of allogeneic organ transplantation.
4. Major surgery, active ulceration, or incomplete wound healing within 1 month prior to the first administration of the study drug (excluding central venous catheter placement, tumor biopsy, or nasogastric tube insertion).
5. Planned elective surgery during the study period.
6. Blood product transfusion or administration of hematopoietic colony-stimulating growth factors (e.g., G-CSF, GM-CSF, M-CSF) within 14 days prior to the first dose of the study drug.
7. Live-attenuated vaccine administration within 30 days prior to the first dose of the study drug.
8. Use of immunosuppressive medications within 14 days prior to the first dose. Exceptions include:

   * Topical, inhaled, or intra-articular corticosteroids.
   * Systemic corticosteroid doses ≤10 mg/day of prednisone or equivalent.
   * Prophylactic corticosteroid use for hypersensitivity reactions (e.g., premedication for CT scans).
9. Active autoimmune or inflammatory diseases, or a history thereof, including inflammatory bowel disease (e.g., colitis, Crohn's disease), diverticulitis (excluding diverticulosis), systemic lupus erythematosus, sarcoidosis, Wegener's syndrome, granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, or uveitis. Exceptions include:

   * Vitiligo or alopecia.
   * Stable hypothyroidism managed with hormone replacement (e.g., post-Hashimoto's thyroiditis).
   * Chronic skin conditions not requiring systemic therapy.
   * Celiac disease controlled by diet.
   * Patients with no active disease within the past 5 years, after consultation with the study investigator.
10. Uncontrolled medical conditions, including but not limited to: persistent or active infections (other than HBV or HCV), symptomatic congestive heart failure, uncontrolled diabetes, uncontrolled hypertension, unstable angina, uncontrolled arrhythmias, active interstitial lung disease, severe chronic gastrointestinal diseases with diarrhea, or psychiatric/social conditions that may limit adherence to study requirements, increase the risk of adverse events (AEs), or impair the ability to provide written informed consent.
11. History of severe bleeding tendency or coagulopathy; clinically significant bleeding symptoms (e.g., gastrointestinal bleeding, hemoptysis) within 1 month prior to the first dose; or ongoing anticoagulation therapy within 10 days prior to the first dose.
12. Arterial thromboembolic events within 6 months prior to the first dose, or venous thromboembolic events graded ≥Grade 3 per NCI CTCAE v5.0.
13. History of another primary malignancy, except:

    * Malignancies treated with curative intent, with no evidence of active disease ≥5 years prior to the first dose and a low risk of recurrence.
    * Non-melanoma skin cancer or malignant melanocytic nevi with no evidence of disease.
    * In situ carcinoma fully treated and with no evidence of disease.
14. Active primary immunodeficiency.
15. Active infections, including tuberculosis or human immunodeficiency virus (HIV 1/2 antibody positivity).
16. Known hypersensitivity or allergic reaction to any component of the study drug or its excipients.
17. Participation in another interventional clinical trial within 1 month prior to the first dose of the study drug.
18. Thromboembolic events (arterial or venous) within 6 months prior to the first dose, such as cerebrovascular accident (including transient ischemic attack, cerebral hemorrhage, or cerebral infarction), deep vein thrombosis, or pulmonary embolism.
19. Participants or their partners who are pregnant or planning pregnancy, or participants who are breastfeeding.
20. Concomitant illnesses deemed by the investigator to pose a significant risk to participant safety or interfere with study completion (e.g., severe diabetes).
21. Other conditions deemed by the investigator to disqualify the participant from study enrollment.

Conversion Success Criteria for Surgical Eligibility

After evaluation by a surgeon, participants meeting the following criteria are considered to have achieved conversion success and are eligible for surgical treatment:

* ECOG performance status ≤1.
* No extrahepatic lesions, or extrahepatic lesions deemed resectable, with no new lesions identified during treatment.
* Tumor vascular occlusion reduced to branch vessels.
* Residual liver volume ≥40% in patients with cirrhosis or ≥30% in patients without cirrhosis after R0 resection.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-05-25 (Estimated); Primary Completion 2026-04-25 (Estimated); Study Completion 2027-04-25 (Estimated)

PRIMARY OUTCOMES:
surgical conversion success rate | From the start of conversion therapy until surgical evaluation or resection, or until it is determined that surgical resection is not feasible.
  Surgical conversion success rate refers to the percentage of subjects who achieve relief after treatment and undergo surgical treatment among the evaluable cases, while also calculating the R0 resection rate and the relief situation based on postoperative pathology.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality
  - Tianjin Cancer Hospital Airport Hospital, Tianjin, Tianjin Municipality